CLINICAL TRIAL: NCT01044628
Title: Multi-Center Randomized Placebo-controlled Trial of Nocturnal Oxygen Therapy in Chronic Obstructive Pulmonary Disease. The International Nocturnal Oxygen (INOX) Trial
Brief Title: The International Nocturnal Oxygen (INOX) Trial
Acronym: INOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Yves Lacasse, Professeur, Laval University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MCT-99512
Record Dates: First submitted 2010-01-06; First posted 2010-01-08 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Nocturnal Desaturation
Keywords: COPD; Oxygen therapy; Nocturnal; Desaturation; INOX
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nocturnal oxygen therapy (N-O2) (Experimental): Oxygen will be delivered overnight to the patients to allow their oxygen saturation to be >90%
  Interventions: Device: Concentrator
- Sham concentrator (Sham Comparator): Sham therapy with ambient air will be given to the patients at night
  Interventions: Device: Sham concentrator

INTERVENTIONS:
Device: Concentrator — Patients allocated to the study group will receive oxygen overnight from an electrically-powered oxygen concentrator (NewLife Intensity Oxygen Concentrator, AirSep Corporation, Buffalo, NY, USA), to allow the oxygen saturation to be >90%
  Arms: Nocturnal oxygen therapy (N-O2)
Device: Sham concentrator — Patients allocated to the control group will receive ambient air delivered overnight through an electrically-powered oxygen concentrator (NewLife Intensity Oxygen Concentrator, Airsep Corporation, Buffalo, NY, USA) rendered ineffective by bypassing the sieve beds. The ineffective concentrators will have the same external appearance as the effective ones, allowing the trial to be double-blinded. We have requested approval by Health Canada in order to proceed with the modifications on the oxygen concentrators. Written permission is pending.
  Arms: Sham concentrator

SUMMARY:
This multicenter randomized placebo controlled trial aims to determine if in patients with COPD not qualifying for LTOT but presenting significant nocturnal arterial oxygen desaturation, whether nocturnal oxygen therapy provided for a period of 4 years decreases mortality or delay the prescription of LTOT.

DETAILED DESCRIPTION:
Background Long-term oxygen therapy (LTOT) is the only component of the management of chronic obstructive pulmonary disease (COPD) that improves survival in patients with severe daytime hypoxemia (defined as an arterial oxygen pressure [PaO2] measured in stable state <= 55 mmHg or in the range 56-59 mmHg when clinical evidence of pulmonary hypertension or polycythemia are noted). In Canada, LTOT is usually provided by a stationary oxygen concentrator and is recommended to be used for at least 15-18 hours a day. Several studies have demonstrated a deterioration in arterial blood gas pressures and oxygen saturation during sleep in patients with COPD. Sleep-related oxygen desaturation often occurs in patients not qualifying for LTOT. The suggestion has been made that the natural progression of COPD to its end stages of chronic pulmonary hypertension, severe hypoxemia, right heart failure, and death is dependent upon the severity of desaturation occurring during sleep. This is an attractive hypothesis and is supported by the fact that hypoxemic episodes during sleep are accompanied by substantial increases in pulmonary arterial pressure and often by important cardiac arrhythmias. Supplemental nocturnal oxygen alleviates both the acute increases in pulmonary arterial pressure and the cardiac arrhythmias. It has been suggested that, over the long run, nocturnal oxygen therapy (N-O2) may halt the progression of long-standing cor pulmonale and prolong survival. Probably due to the fact that the recommendations of scientific societies regarding the indications for and use of N-O2 in COPD not qualifying for conventional LTOT are presently imprecise, a number of patients are currently treated with N-O2 although the beneficial effects of this therapy have not been confirmed.

Objectives Primary objective: To determine, in patients with COPD not qualifying for LTOT but who present significant nocturnal arterial oxygen desaturation, whether N-O2 provided for a period of 4 years decreases mortality or delay the prescription of LTOT.

Secondary objectives: To estimate, in the same population, the cost-utility ratio of nocturnal oxygen therapy over a 4-year period.

Hypotheses In patients with COPD not qualifying for LTOT but who present significant nocturnal arterial oxygen desaturation, N-O2 provided for a period of 4 years is effective in decreasing mortality or delaying the requirement for LTOT; and is cost-effective and favorably compares to other medical interventions.

Research plan Study design: We propose a 4-year, multi-center, placebo-controlled, randomized trial of nocturnal oxygen therapy added to usual care in patients presenting sleep-related oxygen desaturation who do not qualify for LTOT.

Inclusion criteria: (1) patients with a diagnosis of COPD supported by an history of past smoking and obstructive disease with FEV1/FVC < 70%; (2) presence of mild-to-moderate daytime hypoxemia with a daytime PaO2 in the range of 56-69 mmHg; (3) patients fulfilling our definition of nocturnal oxygen desaturation: >= 30% of the recording time with transcutaneous arterial oxygen saturation < 90% on two consecutive recordings.

Intervention:

Nocturnal oxygen therapy: N-O2 will be delivered overnight to allow the oxygen saturation to be > 90%.

Placebo: The patients allocated in the control group will receive room air delivered by defective concentrator. The comparison will be double blind.

Primary outcomes The primary outcomes of this trial are mortality from all cause or requirement for LTOT (composite outcome).

Secondary outcomes Secondary outcomes will include quality of life and utility measures, costs from a societal perspective and compliance with oxygen therapy. Trial duration: The follow-up period lasts at least 4 years. We expect this trial to be completed within 8 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of COPD supported by a history of past smoking and obstructive disease: FEV1<70% predicted, FEV1/FVC<70% and a total lung capacity by body plethysmography >80% predicted;
* Stable COPD at study entry, as demonstrated by (1) no acute exacerbation and (2) no change in medications for at least 6 weeks before enrollment in the trial;
* Non-smoking patients for at least 6 months before enrollment in the trial;
* SpO2 at rest < 95%;
* Patients fulfilling the current definition of nocturnal oxygen desaturation, i.e., >=30% of the recording time with transcutaneous arterial oxygen saturation <90% on at least one of two consecutive recordings;
* Ability ot give informed consent.

Exclusion Criteria:

* Patients with severe hypoxemia fulfilling the usual criteria for continuous oxygen therapy at study entry: PaO2 <=55 mmHg; or PaO2 <= 59 mmHg with clinical evidence of at least one of the following: (1) with right ventricular hypertrophy (P pulmonale on ECG:3 mm leads ll, lll, aVf); (2) right ventricular hypertrophy; (3)Peripheral edema (cor pulmonale); (4) hematocrit >=55%;
* Patients with proven sleep apnea (defined by an apnea/hypopnea index of >=15 events/hour) or suspected sleep apnea on oximetry tracings;
* Patients currently using nocturnal oxygen therapy;
* Patients with known left heart or congenital heart diseases, interstitial lung diseases, bronchiectasis as the main cause of obstructive disease, lung carcinoma, severe obesity (body mass index >= 40 kg/m²), or any other disease that could influence survival.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2010-10; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Composite outcome: all-cause mortality or requirement for continuous oxygen therapy | From date of randomization until the date of prescription of continuous oxygen or date of death from any cause, whichever came first, assessed up to 48 months
  Proportion of patients who died (from any cause) OR required continuous oxygen therapy

SECONDARY OUTCOMES:
Disease-specific quality of life | 48 months
  St-George's respiratory questionnaire; 3 domains analyzed separately : (1) symptoms; (2) activity; (3) impact. Score range for each domain: 0 - 100%; summary score: 0% (perfect health) to 100% (worst).
Generic quality of life | 48 months
  Medical Outcome Survey - Short Form 36 (SF-36); 8 domains analyzed separately: (1) Physical functioning; (2) Role - physical; (3) Bodily pain; (4) General health perception; (5) Energy/vitality ; (6) Social functioning; (7) Role - emotions; (8) Mental health. Domain score and overall score: 0 to 100. Higher score = better health.
Health economics | 48 months
  Costs and health care utilization

CONTACTS AND LOCATIONS:
Overall Officials: Yves Lacasse, MD, MSc, Principal Investigator — Laval University
Locations (28):
- Canada (15):
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - St-Boniface General Hospital, Winnipeg, Manitoba
  - Hôpital Dr Georges-L. Dumont, Moncton, New Brunswick
  - Kingston General Hospital, Kingston, Ontario
  - The Ottawa Hospital (General Campus), Ottawa, Ontario
  - Centre de la santé et des services sociaux de Laval (Cité de la Santé de Laval), Laval, Quebec
  - Hôtel-Dieu de Lévis, Lévis, Quebec
  - Montreal Chest Institute, Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
  - Centre Hospitalier Mount-Sinai, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec (IUCPQ), Québec, Quebec
  - Hôpital régional de Saint-Jérôme, Saint-Jérôme, Quebec
  - CHUS, Fleurimont, Sherbrooke, Quebec
  - Centre de recherche Pneumomédic inc., Trois-Rivières, Quebec
- France (3):
  - Hôpital Nord de Marseille, Marseille
  - Groupe Hospitalier Pitié - Salpêtrière, Paris
  - CHU de Poitiers, Poitiers
- Portugal (6):
  - Centro Hospitalar do Barlavento Algarvio - EPE, Portimão, Algarve
  - Centro Hospitalar de Coimbra, Coimbra
  - Centro Hospitalar da Cova da Beira, Covilha
  - Hospital Pulido Valente - Centro Hospitalar Lisboa Norte, Lisbon
  - Hospital Pedro Hispano Unidade Local de Saude de Matosinhos, Matosinhos Municipality
  - Centro Hospitalara Vila Nova de Gaia-Espinho EPE, Vila Nova de Gaia
- Spain (4):
  - Hospital Galdakao-Usansolo, Galdakao, Biskaia
  - Hospital Universitario de Getafe, Getafe
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Txagorritxu, Vitoria-Gasteiz

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lacasse Y, Series F, Martin S, Maltais F. Nocturnal oxygen therapy in patients with chronic obstructive pulmonary disease: a survey of Canadian respirologists. Can Respir J. 2007 Sep;14(6):343-8. doi: 10.1155/2007/487831. PMID 17885694
- [Derived] Lacasse Y, Series F, Corbeil F, Baltzan M, Paradis B, Simao P, Abad Fernandez A, Esteban C, Guimaraes M, Bourbeau J, Aaron SD, Bernard S, Maltais F; INOX Trial Group. Randomized Trial of Nocturnal Oxygen in Chronic Obstructive Pulmonary Disease. N Engl J Med. 2020 Sep 17;383(12):1129-1138. doi: 10.1056/NEJMoa2013219. PMID 32937046
- [Derived] Lacasse Y, Bernard S, Series F, Nguyen VH, Bourbeau J, Aaron S, Maltais F; International Nocturnal Oxygen (INOX) Research Group. Multi-center, randomized, placebo-controlled trial of nocturnal oxygen therapy in chronic obstructive pulmonary disease: a study protocol for the INOX trial. BMC Pulm Med. 2017 Jan 9;17(1):8. doi: 10.1186/s12890-016-0343-9. PMID 28069009

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-10-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT01044628/Prot_SAP_000.pdf